CLINICAL TRIAL: NCT06587828
Title: A Biospecimen Collection Study to Identify the Targets of Disease-Reactive T Cells in Patients With Autoimmune Disease
Status: Recruiting | Type: Observational
Sponsor: TScan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-05
Record Dates: First submitted 2024-04-18; First posted 2024-09-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Diseases; Ulcerative Colitis; Multiple Sclerosis; Scleroderma; Ankylosing Spondylitis; Celiac Disease; Non-radiographic Axial Spondyloarthritis (Nr-axSpA); Crohn&Amp;#39;s Disease; Birdshot Chorioretinitis
Keywords: Autoimmune Diseases; Multiple Sclerosis; Systemic Sclerosis; Ankylosing Spondylitis; Scleroderma; Inflammatory Bowel Disease; Crohn's Disease; Non-radiographic axial spondyloarthritis (nr-axSpA); Birdshot Chorioretinitis
MeSH Terms: conditions — Autoimmune Diseases; Colitis, Ulcerative; Multiple Sclerosis; Scleroderma, Diffuse; Spondylitis, Ankylosing; Celiac Disease; Non-Radiographic Axial Spondyloarthritis; Birdshot Chorioretinopathy; Scleroderma, Systemic; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Crohn's Disease and Ulcerative Colitis: Mucosal tissue from inflamed colon, rectum or ileum and healthy colon tissue and blood. Celiac Disease: Small intestine tissue and blood. Ankylosing Spondylitis: synovial fluid and blood. Multiple Sclerosis: Cerebrospinal fluid and blood. Scleroderma: Skin tissue and blood. Systemic Sclerosis: Inflamed lung tissue and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Inflammatory Bowel Diseases- Crohn's Disease and Ulcerative Colitis: Group A: IBD-Treatment Naïve Crohn's: Patients that are scheduled to have an endoscopic procedure to confirm a suspected diagnosis of Crohn's disease and are not currently on any Crohn's directed treatment.
  Group B: IBD-On-Treatment Crohn's: Patients with an established diagnosis of Crohn's disease and are only on treatments that are allowed under this protocol (see Inclusion and Exclusion criteria) and consent to have extra biopsies obtained from inflamed and normal colon for research purposes during a planned endoscopy for their standard clinical care.
  Group C: IBD-Ulcerative Colitis: Patients with established or suspected diagnosis of ulcerative colitis who may be on treatments that are allowed under this protocol (see Inclusion and Exclusion criteria).
  Interventions: Companion blood samples with colonoscopy and biopsies for participants with Crohn's Disease or Ulcerative Colitis
  Interventions: Procedure: Companion blood samples with procedure
- Celiac Disease: Small intestine endoscopic biopsies obtained during endoscopy: Group A Celiac Disease: Excess small intestine biopsies obtained during endoscopy from patients with celiac disease or from patients who are suspected to have celiac disease. A companion blood sample will be drawn on or around the same day.
  Group B Celiac Disease: Patients who are suspected to have celiac disease or are known to have celiac disease and who undergo a research endoscopy of the small intestine to obtain biopsy samples from the small intestine. A companion blood sample will be drawn on or around the same day.
  Interventions: Companion blood samples with upper endoscopy and biopsies.
  Interventions: Procedure: Companion blood samples with procedure
- Ankylosing spondylitis or non-radiographic axial spondyloarthritis (nr-axSpA) (HLA-B27 positive): Group A ankylosing spondylitis- arthrocentesis: HLA-B27 positive patients with known or suspected ankylosing spondylitis or nr-axSpA with inflammatory joint involvement who consent to arthrocentesis done for research purposes. A blood sample drawn on or around the same day of the procedure is also required. A minimum of 2 mL and up to 10 mL of joint aspiration fluid is required.
  Group B ankylosing spondylitis- surgery: HLA-B27 positive patients with known or suspected ankylosing spondylitis or nr-axSpA planned for surgery for their standard clinical care who consent to have excess materials from their resected joint tissues used for research purposes. Bone, joint or biologic materials from the surgical resection is acceptable. A blood sample drawn on or around the same day of the procedure is also required.
  Interventions: Companion blood samples with arthrocentesis
  Interventions: Procedure: Companion blood samples with procedure
- Multiple Sclerosis. Excess CSF collected during lumbar puncture: A. Multiple Sclerosis Group A: Extra CSF from standard clinical procedure in patients diagnosed with multiple sclerosis and have a planned lumbar puncture for standard clinical care where extra CSF may be obtained for standard of care. A blood sample drawn on or around the same day is required. CSF in excess of clinical laboratory requirements will be used for study purposes. 2 mL to 10 mL of CSF is required. Up to 20 patients will be recruited into research procedure group.
  B. Multiple Sclerosis Group B: Research CSF collection - Patients will have CSF collected during a lumbar puncture that is not required for standard clinical care and will also have a companion blood sample collected. The patient will consent to a research lumbar puncture and will be enrolled into the research CSF collection cohort. 2 mL to 10 mL of CSF is required. Up to 10 patients will be recruited into this group.
  Interventions: Companion blood samples with lumbar puncture
  Interventions: Procedure: Companion blood samples with procedure
- Scleroderma. Skin tissue biopsy: A. Scleroderma Group A: Excess Tissue - Excess skin tissue obtained during a planned skin tissue biopsy and with a companion blood sample. A minimum sample of a a single 3 mm punch biopsy is required and up to 3 punch biopsies will be allowed. Up to 10 patients will be recruited into this group.
  B. Scleroderma Group B: Research Skin Biopsy - Patients that agree to a research skin tissue biopsy, not otherwise clinically indicated and obtained at any one point in time, and with a companion blood sample. For skin biopsies, a minimum sample of a single 3 mm punch biopsy is required and up to 3 punch biopsies will be allowed. Up to 10 patients will be recruited into this group.
  Interventions: Companion blood samples with skin biopsy
  Interventions: Procedure: Companion blood samples with procedure
- Systemic Sclerosis with pulmonary involvement: Patients would consent to have excess materials from their bronchoscopy, bronchoalveolar lavage fluid or thoracoscopy done for standard of care purposes. Patients should not undergo these procedures unless required for standard clinical care. There is no minimum tissue requirement for this cohort. Up to 10 patients will be recruited into this group.
  Interventions: Companion blood samples with biopsy
  Interventions: Procedure: Companion blood samples with procedure
- Other Autoimmune Disease such as psoriasis, vitiligo, type 1 diabetes and others: A. Other Autoimmune Group A: Excess Biologic Material - Excess material sourced from a part of the body exhibiting clinical symptoms of autoimmune disease +/- nearby normal biologic materials, and with a companion blood sample. While there is no minimum tissue requirement for this cohort, tissue requirements from other autoimmune diseases described above may be used to guide tissue collection sample amounts.
  B. Other Autoimmune Group B: Research Biologic Material - Research skin tissue biopsy, other tissue biopsy or biologic materials collected from an affected part of the body +/- normal healthy biologic materials, and with a companion blood sample. In the instance of a skin biopsy, a minimum of a single 3 mm punch biopsies, and up to three, 3 mm punch biopsies, will be obtained.
  Interventions: Procedure: Companion blood samples with procedure
- Evolving autoimmune disease: Serial sampling of excess materials, with companion blood samples, can be obtained at intervals consistent with excess materials collected for clinical care.
  Interventions: Procedure: Companion blood samples with procedure
- Previously cryopreserved, dissociated tissue obtained from a biobank or tissue repository: These samples will have been collected from patients with autoimmune diseases, at any one time point after diagnosis and with a companion blood sample.
  Interventions: Procedure: Companion blood samples with procedure

INTERVENTIONS:
Procedure: Companion blood samples with procedure — Participants in all cohorts will have a companion blood sample obtained on or around the time of the procedure intended to obtain tissue or fluid.

SUMMARY:
The most clinically meaningful way to discover new targets of T cells in autoimmune diseases is to study the tissues of patients with active autoimmune disease mediated organ inflammation. These tissues contain both cytotoxic and helper T cells that are driving their disease, and these T cells are being guided by TCRs that recognize tissue-specific targets. By collecting tissue when a patient has active inflammation, it is possible to determine which T cells are activated and undergoing clonal expansion in the patient's diseased organ. TScan has developed a genome-wide, high-throughput technology to determine the natural, physiological target of any TCR (Kula, 2019). The goal of this study is to isolate T cells from inflamed tissues and matched blood samples and/or matched normal tissues (for patients with inflammatory bowel diseases). T cell clones that are expanded in diseased tissues relative to blood or normal tissues will be selected and the targets of their TCRs will be defined using TScan's genome-wide, high-throughput target ID technology.

The goal of this study is to discover a collection of peptide targets, along with their associated TCRs to be developed as new tolerogenic therapies for patients with autoimmune diseases.

ELIGIBILITY:
Cohort Legend: Cohort 1: Inflammatory Bowel Diseases - Crohn's Disease or Ulcerative Colitis, Cohort 2: Celiac Disease, Cohort 3: Ankylosing spondylitis or non-radiographic axial spondyloarthritis (nr-axSpA), Cohort 4: Multiple Sclerosis, Cohort 5: Scleroderma, Cohort 6: Systemic Sclerosis with pulmonary involvement, Cohort 7: Other Autoimmune Disease, Cohort 8: Apparent Evolving Autoimmune Disease, Cohort 9: Frozen Cryopreserved

Inclusion Criteria:

* Study cohorts 1,2,3,4,5,6,7,8.9: Known or suspected diagnosis, with subsequent diagnostic confirmation, of one of the following cohorts associated with the following autoimmune diseases:
* Inflammatory Bowel Diseases - Crohn's Disease or ulcerative colitis
* Celiac disease
* Ankylosing spondylitis or Non radiographic axial spondyloarthritis (nr-axSpA)
* Multiple sclerosis
* Scleroderma
* Systemic sclerosis with pulmonary involvement
* Other autoimmune disease (as agreed between Investigator and Sponsor)
* Apparent evolving autoimmune disease
* Frozen cryopreserved
* Age equal or greater than 18 years at time of informed consent.
* Ability to understand and willingness to sign an informed consent document when informed consent is required by an ethical review board.
* On disease-modifying treatments that are not known to be directly T cell toxic.

Such treatments are allowed and include:

* Non-steroidal anti-inflammatory drugs including aspirin, ibuprofen, acetaminophen, celecoxib, indomethacin, diclofenac, etodolac, naproxen, meloxicam, sulindac, nabumetone amongst others.
* Tumor necrosis factor alpha (TNF-alpha) antagonists including infliximab (Remicade), adalimumab (Humira), certolizumab pegol (Cimzia), etanercept (Enbrel), golimumab (Simponi) and biosimilar drugs with the same generic name.
* Interleukin-12/23 antagonists including ustekinumab (Stelara) and risankizumab-rzaa (Skyrizi)
* Alpha-4-integrin antagonists including vedolizumab (Entyvio), natalizumab (Tysabri)
* Interleukin-17 inhibitors including secukinumab (Cosentyx), ixekizumab (Taltz)
* Recombinant interferon beta
* CD20 antagonists including rituximab (Rituxan), ocrelizumab (Ocrevus), ofatumumab (Kesimpta)
* Oral fumarates including dimethyl fumarate (Tecfidera), diroximel fumarate (Vumerity), monomethyl fumarate (Bafiertam)
* Oral sphingosine 1-phosphate receptor (S1PR) modulators including fingolimod (Gilenya), siponimod (Mayzent), ozanimod (Zeposia), ponesimod (Ponvory)
* Oral glatiramer acetate (copolymer 1; Copaxone)
* Patient is an appropriate candidate for a procedure to obtain a biopsy, tissue samples or biologic materials during a clinically indicated procedure where it is expected that excess materials could be used for research OR
* In the opinion of the clinical investigator, a patient is an appropriate, low-risk candidate for a research only procedure to obtain a biopsy, tissue samples or biologic materials.

Exclusion Criteria:

* On treatment with drugs that are known to be T cell toxic and cannot be held for at least 4 weeks or longer. The following treatments are not allowed except in designated cohorts when approved by Sponsor:
* Glucocorticoids including prednisone, methylprednisolone (Solu-medrol), budesonide (Entocort), hydrocortisone (Solu-cortef), dexamethasone (Decadron), betamethasone (Betaject)
* Sulfasalazine (Azulfidine)
* Aminosalicylates including mesalamine/ mesalazine (Asacol, Pentasa).
* Thiopurines including azathioprine (Imuran) and 6-mercaptopurine (Purixan)
* Systemic JAK inhibitors including tofacitinib (Xeljanz), abrocitinib (Cibinqo), baricitinib (Olumiant), upadacitinib (Rinvoq)
* CD52 inhibitors including alemtuzumab (Campath)
* Methotrexate
* Cladribine
* Teriflunomide (Aubagio)
* Concurrent disease or condition that would make the patient inappropriate for study participation, or any serious medical or psychiatric disorder that would interfere with the subject's safety.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Patients receiving research biopsy procedures will not have a history of serious or life-threatening allergic reaction to local anesthetics (i.e., lidocaine, xylocaine), if local anesthetic is required for the procedure or to medications used for sedation during a procedure.
* Pregnant or nursing women are excluded because there may be unanticipated adverse events and increased risk to both mother and fetus in the setting of local anesthetic or study procedures.
* Any other medical or psychiatric condition, which in the opinion of the patient's treating clinician, would make participation in this protocol unreasonably hazardous for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a known or suspected autoimmune disease will be enrolled into the study. Additionally, patients who have an apparent evolving autoimmune disease may be eligible.
  Patients with autoimmune disease who had excess materials cryopreserved in a manner that is expected to yield sufficient T cells for this research study, and where biologic samples were ethically obtained, will be utilized for this study.
  Both men and women and members of all races and ethnic groups are eligible for this protocol. It is expected that the mix of patients entering this study will reflect the demographics of the clinic population seen in hospitals and associated clinics in the region from which the biologic materials are collected.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Identify peptide targets together with their associated TCRs in patients with autoimmune diseases under study. | 3 Years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Knowledge Research Center, Orange, California
  - Cura Clinical Research, Sherman Oaks, California
  - Arnold Arthritis & Rheumatology, Skokie, Illinois
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Massachusetts Eye Research and Surgery Institution (MERSI), Waltham, Massachusetts
  - Susquehanna Research Group, Harrisburg, Pennsylvania
  - Nexus Research, Cranston, Rhode Island
  - RI Rheumatology, Cranston, Rhode Island
  - Palmetto Gastroenterology Clinical Research, LLC, Summerville, South Carolina
  - Novel Research, Bellaire, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin